CLINICAL TRIAL: NCT05050240
Title: Identification of Brown Fat-derived Blood-borne Factors as Biomarkers of Metabolic Health in Humans
Brief Title: BATokines as Biomarkers of Brown Fat in Humans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KPL-1023
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Healthy Lifestyle
Keywords: metabolism; cold exposure; brown fat; blood biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Exposure (Experimental): The cold vest procedure: The first blood draw will be taken from participants before the cooling procedure (time 0, 30mL blood). Participants will then be requested to put on hospital scrubs and the cooling vest will be placed on them. Since muscle shivering is an alternative way of heat production (skeletal thermogenesis), we will first determine individual 'shivering threshold' for each participant (coldest tolerable temperature; typically 14°C / 57.2F), based on participant-report and direct observation. The cold vest will then be kept on for 3 hours with a temp set to the coldest tolerable temperature (shivering threshold +2°C (~16-17°C / 60.8F-62.6F) and body temperature will be monitored by a tympanic thermometer. Following 3 hours, 30mL of blood will be drawn (Time 180min). All participants will be re-warmed with blankets after cooling has been completed, and offered a warm drink and a snack.
  Interventions: Other: Cooling Vest Procedure
- Fasted procedure without cooling (Active Comparator): This arm has been added in order to exclude the effects of prolonged fasting on blood analytes. Previously enrolled participants will be re-invited to donate blood after 12hr fast and 3hrs later (15hr fast) without the cooling procedure. Participants will be re-consented for this lab appointment. The night prior the visit, the participants will be instructed to fast from 10:00pm. At the time of visit vital signs and anthropomorphic measurements will be taken.
  Blood Draw: The first blood draw will take place in the morning. Participant will then be asked to sit in the procedure room for 3 hours at room temperature; second blood draw will take place after 3 hrs. Total of 38ml of blood will be drawn. Blood will be used for clinical labs (fasting glucose, Hba1c, TSH, TG) and research.
  Interventions: Other: Fasting overnight

INTERVENTIONS:
Other: Cooling Vest Procedure — A cold vest will be placed on the participant (consisting of a water-perfused CFA wearable vest, size S-M or M-L with adjustable straps Polar Products, Stow, OH; attached to a small 'cooler' reservoir to circulate cold water between the vest and the cooler; Product link: https://www.polarproducts.com/polarshop/pc/CoolOR-13-Quart-System-with-Arctic-Chiller-p24757.htm This product is safe and recommended by experimental guidelines and BARCIST criteria for human BAT studies. Note, the cooling vest will be cleaned between participants according to the manufacturer's guidelines found here: https://www.polarproducts.com/polarshop/pc/catalog/pdf/Polar_CoolFlow_Manual.pdf.
  Briefly, the vest will be hand washed with a mild detergent and warm soapy water and air-dried. The vest will then be stored in a clean, dry environment with ventilation.
  Arms: Cold Exposure
Other: Fasting overnight — Participants will be requested to refrain from food and caloric drinks overnight (starting at 10pm) prior to the hospital visit. Blood will then be drawn the following morning (between 8 and 9am) and 3hrs later (between 11am and noon). Participants will be sat in a room with ambient temperature (room temperature w/o cooling) between the two blood draws.
  Arms: Fasted procedure without cooling

SUMMARY:
Brown adipose tissue (BAT) burns excess calories to produce heat in response to environmental cold. Rapidly growing evidence from rodent and human studies suggests that the presence and activation of brown fat are far more beneficial for whole body metabolism and cardiometabolic health than previously appreciated. Despite the clear associations between brown fat and metabolic health, we lack both: cost-effective means of detecting brown fat in humans as well as comprehensive insights into how brown fat facilitates metabolism on a molecular level in humans.

Emerging evidence suggests that the benefits of brown fat activation are mediated, at least in part, by secretion of specific molecules into the bloodstream which signal to metabolically active organs such as skeletal muscle, liver and brain. A number of these so-called brown adipokines (or BATokines) have now been discovered in mice and shown to positively impact glucose homeostasis, liver and muscle function. Human deep-neck brown fat biopsies reveal that >1000 molecules could potentially be secreted from brown fat, and >400 are released by human brown fat cells in a dish, representing a major opportunity for discovery of high translational value.

Here, we aim to identify a screen of first potential blood biomarkers of brown fat in healthy young humans. This will be achieved by analyzing plasma proteins in subjects with 'inactive brown fat' (warm) and 'activated brown fat' (3-hr cold exposure, cooling vests) using high-throughput technologies (SOMAscan and O-link) to identify temperature-sensitive brown fat-enriched molecules. This preliminary data will guide a larger follow up study in which we envision studying lean and obese (insulin sensitive and insulin resistant) subjects of various age groups and race/ethnicity. Human BATokines identified here will become primary targets for manipulation in experimental animals to assess their therapeutic potential against obesity, T2D, and associated diseases. Additionally, since current methods of brown fat detection in human rely on deep neck biopsies or costly 18-FDG-PET/CT scans, identification of blood biomarkers of brown fat would offer a cost-effective and non-invasive alternative for prediction of metabolic health in humans.

DETAILED DESCRIPTION:
Fat plays a fundamental role in regulating metabolic health due to its capacity to store excess calories (white adipose tissue; WAT) or burn them to produce heat (brown adipose tissue, BAT). While white fat cells are located in deposits beneath the skin (subcutaneous) or around the internal organs (visceral) and expand with obesity, brown fat cells reside predominantly in the deep neck area and have evolved to turn fuel into heat (a process termed thermogenesis) when activated by environmental cold. This calorie-burning property of BAT suggest it is a type of 'good fat' which may protect us from conditions such as obesity. A wealth of mouse data confirms that activation of BAT via cold exposure provides significant health benefits to experimental animals, including protection from diet-induced obesity and improved glucose metabolism. BAT has only recently been detected in adult humans, which has led to efforts to understand its physiology and investigate whether its activity can be manipulated to treat metabolic diseases. Notably, in addition to storing or burning fat, adipose tissue secretes a large number of hormone-like factors into the bloodstream, known to affect blood glucose levels and insulin sensitivity (adiponectin, adipsin) as well as appetite and energy expenditure (leptin). Although many such factors have been identified in white fat, little is known about the proteins secreted from brown fat, particularly in humans.

In a recent study of 52,000 patients with 18-FDG-PET/CT scans to identify the presence of brown fat, we found that BAT+ individuals had significantly reduced odds of type 2 diabetes (T2D), coronary artery disease, and congestive heart failure, compared to matched individuals who did not have brown fat. A smaller independent study demonstrated that short-term activation of BAT with cooling jackets significantly improved insulin sensitivity in T2D patients. These findings collectively reveal that BAT carries extraordinary potential to impact metabolic health in humans.

Metabolic benefits linked with BAT cannot be explained by the generation of heat (thermogenesis) alone. Emerging evidence suggests that BAT secretes specific molecules into the bloodstream. A number of these so-called brown adipokines (or BATokines) have now been discovered in mice and shown to positively impact whole body glucose metabolism and liver function, reducing the susceptibility to metabolic disease. However, the 'secretome' of brown fat has not been well studied in humans, and hence the relevance of these BATokines to our physiology remains unclear. In support of this unexplored research avenue, gene expression data from deep-neck BAT biopsies reveal that >1,000 molecules could potentially be secreted from BAT in humans, and 431 were identified as being released from human BAT cells in a dish, but a comprehensive validation of these proteins in blood samples of participants with activated BAT is lacking.

The aim of this study is to identify a panel of plasma proteins induced by activation of brown fat in young healthy human participants and provide pilot data for a larger biomarker study. We will employ novel unbiased multiplex tools to identify up to 7,000 unique proteins of various abundances, in subjects before and after cooling. Using these data, we will be able to identify common circulating factors that correlate with BAT activation, and subsequently compare them with pre-existing gene expression data to find polypeptides secreted, shedded or otherwise released specifically by BAT. While this study will focus on the identification of proteins, we also have the potential to survey small molecule metabolites secreted into the circulation. This list of BATokines will become instrumental for validation and retro-translation of mouse data from our lab and the larger scientific community interested in the metabolic benefits conveyed by BAT. In addition to the discovery of potential therapeutic targets, the blood screen may become a valuable data platform for clinical biomarkers of brown fat. Since current methods of BAT detection in human rely on deep neck biopsies and/or costly 18-FDG-PET/CT scans, identification of blood factors that circulate proportionally to BAT activity or correlate with the presence or amount of BAT would offer a cost-effective, non-invasive alternative in human participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 28
* BMI >19 and < 25

Exclusion Criteria:

* Diabetes type I or II (self-report)
* Diagnosis of thyroid disease (including goiter, hyperthyroidism, hypothyroidism, thyroiditis) (self-report)
* Diagnosis with cancer including skin cancer (self-report)
* Diagnosis or evidence of Raynaud's Syndrome or systemic sclerosis (self report)
* Previously or currently diagnosed with SARS-Cov-2 infection/COVID-19 (secondary to unknown immune responses)
* Any vaccine administration within two weeks preceding the study procedure
* Currently pregnant
* Currently taking any prescribed medication other than oral contraceptives
* Treatments for weight loss or any other supplements that may alter weight or metabolism are not acceptable (vitamins are acceptable)
* Has consumed nicotine (smoking, inhaling, ingesting) within the last within the last 6 months
* Has used illicit drugs within the last 6 months
* Any medical, psychological, or social condition that, in opinion of principle investigators, would jeopardize the health or well-being of the participant during the study procedure or integrity of the data

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of cold-regulated blood proteome | Before and after a 3 hour cooling procedure
  Mass spectrometry generates a list of proteins for each sample. We will compare fold of change before and after cooling - a true change is defined as 1.5-fold.

SECONDARY OUTCOMES:
Changes in HbA1c post cooling procedure using absorbance assay | Before and after a 3 hour cooling procedure
  Absorbance assay
Changes in insulin post cooling procedure using enzyme-linked immunosorbent assay (ELISA) | Before and after a 3 hour cooling procedure
  ELISA
Changes in triglycerides post cooling procedure using absorbance assay | Before and after a 3 hour cooling procedure
  Absorbance assay
Changes in TSH post cooling procedure using absorbance assay | Before and after a 3 hour cooling procedure
  Absorbance assay

CONTACTS AND LOCATIONS:
Overall Officials: Kaja Plucinska, PhD, Principal Investigator — The Rockefeller University; Paul Cohen, PhD, Study Director — The Rockefeller University
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No